CLINICAL TRIAL: NCT05260437
Title: A Phase 1, Open-label, Safety, Reactogenicity, and Immunogenicity Trial of the CV2CoV mRNA Vaccine Against SARS CoV 2 in Seropositive Adult Participants
Brief Title: Safety, Reactogenicity, and Immunogenicity Trial of CV2CoV mRNA Vaccine Against SARS-CoV-2 in Seropositive Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: CureVac (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 217741
Record Dates: First submitted 2022-02-25; First posted 2022-03-02 (Actual); Results first posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-03

CONDITIONS: COVID-19; SARS-CoV-2
Keywords: COVID-19; Pandemic; Booster vaccination
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- CV2CoV Dose Cohort 1 (Group 1a 2μg) (Experimental): Participants received 2 μg CV2CoV intramuscularly.
  Interventions: Biological: CV2CoV (2 µg)
- CV2CoV Dose Cohort 1 (Group 1b 4μg) (Experimental): Participants received 4 μg CV2CoV intramuscularly.
  Interventions: Biological: CV2CoV (4 µg)
- CV2CoV Dose Cohort 2 (8 μg) (Experimental): Participants received 8 μg CV2CoV intramuscularly.
  Interventions: Biological: CV2CoV (8 µg)
- CV2CoV Dose Cohort 3 (12 μg) (Experimental): Participants received 12 μg CV2CoV intramuscularly.
  Interventions: Biological: CV2CoV (12 µg)
- CV2CoV Dose Cohort 4 (16 μg) (Experimental): Participants received 16 μg CV2CoV intramuscularly.
  Interventions: Biological: CV2CoV (16 µg)
- CV2CoV Dose Cohort 5 (20 μg) (Experimental): Participants were scheduled to receive 20 μg CV2CoV Intramuscularly, but there were no participants enrolled in this group, and hence, there was no vaccine administered in this study group.
  Interventions: Biological: CV2CoV (20 µg)

INTERVENTIONS:
Biological: CV2CoV (2 µg) — Study vaccine was administered as a single intramuscular injection.
  Arms: CV2CoV Dose Cohort 1 (Group 1a 2μg)
Biological: CV2CoV (4 µg) — Study vaccine was administered as a single intramuscular injection.
  Arms: CV2CoV Dose Cohort 1 (Group 1b 4μg)
Biological: CV2CoV (8 µg) — Study vaccine was administered as a single intramuscular injection.
  Arms: CV2CoV Dose Cohort 2 (8 μg)
Biological: CV2CoV (12 µg) — Study vaccine was administered as a single intramuscular injection.
  Arms: CV2CoV Dose Cohort 3 (12 μg)
Biological: CV2CoV (16 µg) — Study vaccine was administered as a single intramuscular injection.
  Arms: CV2CoV Dose Cohort 4 (16 μg)
Biological: CV2CoV (20 µg) — Study vaccine was planned to be administered intramuscularly. No vaccine was administered in the CV2CoV (20 µg) Group, since there were no participants enrolled in it.
  Arms: CV2CoV Dose Cohort 5 (20 μg)

SUMMARY:
Prevention of COVID-19 caused by SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

1. Must provide documented informed consent prior to any study procedures being performed.
2. Is capable of understanding and agrees to comply with planned study procedures and to be available for all study visits, including being willing and able to use electronic devices during the study.
3. Has received at least 2 doses of Pfizer-BioNTech (Comirnaty) or Moderna (Spikevax) mRNA COVID-19 vaccine with the last dose of vaccine received at least 6 months prior to Screening and has provided documentation of receiving the vaccination series.
4. Negative for SARS-CoV-2 infection by RT-PCR test at Screening.
5. Is a male or nonpregnant female 18 to <65 years of age (younger adult group) or ≥65 years of age (older adult group) at Screening.
6. Has a body mass index of 18 to 34.9 kg/m^2, inclusive, at Screening.
7. If the participant is a woman of child bearing potential the participant agrees to practice true abstinence or use at least 1 highly effective form of contraception for at least 30 days prior to study vaccination up to 3 months after study vaccination.
8. Agrees to refrain from blood or plasma donation from Screening and throughout the end of the study.
9. Is healthy or medically stable as determined by medical history, clinical laboratory tests, vital sign measurements, and physical examination findings, as determined by investigator judgment.

Exclusion Criteria:

1. Participant is female and has a positive serum pregnancy test result at Screening or plans to become pregnant during the study.
2. Participant is female and is breastfeeding or plans to breastfeed from study vaccination to 3 months after study vaccination.
3. Has any clinically significant abnormal biochemistry or hematology finding (defined as ≥Grade 1) at Screening.
4. Has any medical disease or condition that, in the opinion of the investigator, precludes study participation. This includes any acute, subacute, intermittent, or chronic medical disease or condition that would place the participant at an unacceptable risk of injury, render the participant unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the participant's successful completion of the trial.
5. Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease or immunosuppressive/cytotoxic therapy.
6. History of myocarditis, pericarditis, or idiopathic cardiomyopathy, or presence of any medical condition that increases risk of myocarditis or pericarditis, including cocaine abuse, cardiomyopathy, endomyocardial fibrosis, hypereosinophilic syndrome, hypersensitivity myocarditis, eosinophilic granulomatosis with polyangiitis, persistent myocardial viral infection (eg, due to enterovirus or adenovirus), and celiac disease.
7. Has an acute febrile illness with a temperature ≥38.0°C or ≥100.4°F observed by the participant or at the study site within 72 hours prior to study vaccination. Participants with suspected COVID-19 symptoms should be excluded and referred for medical care.
8. Has a prior confirmed diagnosis of chronic hepatitis B, hepatitis C, or HIV 1/2 infection or evidence of active infection at Screening.
9. Has participated or plans to participate in another investigational study involving any investigational drug or device within 60 days or 5 half-lives, whichever is longer, before study vaccination and throughout the end of the study.
10. Has previously participated in an investigational vaccine study with investigational vaccine administered within 6 months of study vaccination OR has received the last dose of >1 COVID-19 vaccine series (investigational and/or authorized) in the last 12 months.
11. Has received or plans to receive any licensed vaccine within 4 weeks before or after study vaccination. Inactivated vaccines for influenza are permitted during the study if they are administered at least 14 days before or after study vaccination.
12. Is planning to receive a COVID-19 booster vaccination for the duration of the study (for adults who are not covered by local recommendations to receive booster per current standard of care) or is planning to receive a COVID-19 booster vaccination on or before Day 29 of the study (for adults covered by local recommendations to receive booster).
13. Has received or plans to receive immunoglobulins or any blood or blood products within 90 days before study vaccination and throughout the study.
14. Has a history of hypersensitivity or severe allergic reaction, including anaphylaxis, generalized urticaria, angioedema, and other significant reactions to any previous vaccine or any component of the IP.
15. Has a history of hypersensitivity or severe allergic reaction (including anaphylaxis, generalized urticaria, angioedema, and other significant reactions) to beta lactam antibiotics.
16. Reports chronic use (more than 14 continuous days) of any medication that may be associated with changes in immune function including, but not limited to, systemic corticosteroids exceeding 10 mg/day of prednisone equivalent, allergy injections, immunoglobulins, interferons, immunomodulators, cytotoxic drugs, or other similar or toxic drugs within 6 months of study vaccination.
17. Has a bleeding disorder or prior history of significant bleeding or bruising after IM injections or venipuncture.
18. Has a history of alcohol abuse or other recreational drug use (excluding cannabis) within 6 months before study vaccination.
19. Has any abnormal skin condition or permanent body art that would interfere with the ability to observe local reactions at the study vaccination injection site.
20. Has had known close contact with anyone who had a confirmed SARS-CoV-2 infection within 14 days before study vaccination.
21. Participant is an employee or family member of the investigator or study site personnel.
22. Has any self-reported or medically-documented significant medical or psychiatric condition. Significant medical conditions include, but are not limited to, the following:

    1. Moderate or severe respiratory disease
    2. Uncontrolled hypertension, defined as an average systolic blood pressure ≥140 mmHg for participants ≤60 years old, and ≥150 mmHg for participants >60 years old, or a diastolic blood pressure ≥90 mmHg for any age
    3. Significant cardiovascular disease or history of myocarditis or pericarditis
    4. Neurological or neurodevelopmental conditions
    5. Ongoing malignancy or recent diagnosis of malignancy in the last 5 years (excluding basal cell and squamous cell carcinoma of the skin)
    6. Tuberculosis or nontuberculosis mycobacterial infection
    7. Autoimmune disease, including hypothyroidism without a defined nonautoimmune cause
    8. Immunodeficiency of any cause, including from solid organ transplant, blood or bone marrow transplant, use of corticosteroids, or use of other immune weakening medicines
    9. Type 1 or 2 diabetes mellitus regardless of disease control
23. Has any of the following self-reported or medically-documented risk factors for severe COVID-19:

    1. Cancer
    2. Chronic kidney disease
    3. Sickle cell disease
    4. Cerebrovascular disease
    5. Cystic fibrosis
    6. Chronic liver disease
    7. Pulmonary fibrosis
    8. Thalassemia
    9. Smoking or other inhaled substance use, including tobacco, cannabis, or nicotine vapors, with an average of ≥5 cigarettes a day or equivalent (currently or within 1 year of Screening).
24. Has a history of documented SARS-CoV-2 infection or COVID-19 within 6 months before Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Lynn Institute of Denver - ERN, Aurora, Colorado
  - GSK Investigational Site, Hallandale, Florida
  - MD Clinical - Velocity, Hallandale, Florida
  - GSK Investigational Site, Lakeland, Florida
  - Accel Research Sites, Lakeland, Florida
  - GSK Investigational Site, Miami, Florida
  - Suncoast Research Group LLC - ERN-PPDS, Miami, Florida
  - GSK Investigational Site, Palm Springs, Florida
  - Affinity Health Corp, Oak Brook, Illinois
  - GSK Investigational Site, Oak Brook, Illinois
  - GSK Investigational Site, Cleveland, Ohio
  - Velocity Clinical Research - Cleveland, Cleveland, Ohio
  - GSK Investigational Site, Norman, Oklahoma
  - Lynn Institute of Norman - ERN - PPDS, Norman, Oklahoma
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - GSK Investigational Site, Cedar Park, Texas
  - GSK Investigational Site, Dallas, Texas
  - Research Your Health - Elite, Plano, Texas
  - DM Clinical - Cyfair Clinical Research Center, Tomball, Texas
  - GSK Investigational Site, Tomball, Texas
  - GSK Investigational Site, West Jordan, Utah
  - Velocity Clinical Research - Salt Lake City - Jordan Valley-ERN-PPDS, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 13 centers in the United States.
Pre-assignment Details: Escalation to the next higher dose cohorts was based on the Safety Review Team (SRT) review of safety data from the same age group. GlaxoSmithKline Biologicals SA (GSK) and CureVac decided to stop further enrollment or vaccination in the CV2-SARS-CoV-2-002 (217741) dose escalation study. This decision was taken because the data accumulated were considered sufficient to determine next steps in vaccine platform development. Therefore, enrollment in CV2CoV Dose Cohort 5 (20 µg) was never opened.
Groups:
- CV2CoV Dose Cohort 1 (Group 1a 2µg): Participants received 2 µg CV2CoV intramuscularly.
- CV2CoV Dose Cohort 1 (Group 1b 4µg): Participants received 4 µg CV2CoV intramuscularly.
- CV2CoV Dose Cohort 2 (8 µg): Participants received 8 µg CV2CoV intramuscularly.
- CV2CoV Dose Cohort 3 (12 µg): Participants received 12 µg CV2CoV intramuscularly.
- CV2CoV Dose Cohort 4 (16 µg): Participants received 16 µg CV2CoV intramuscularly.
Period: Overall Study
Arm/Group | CV2CoV Dose Cohort 1 (Group 1a 2µg) | CV2CoV Dose Cohort 1 (Group 1b 4µg) | CV2CoV Dose Cohort 2 (8 µg) | CV2CoV Dose Cohort 3 (12 µg) | CV2CoV Dose Cohort 4 (16 µg)
Started | 24 | 23 | 20 | 21 | 11
Completed | 16 | 20 | 15 | 14 | 9
Not Completed | 8 | 3 | 5 | 7 | 2
Not completed — Lost to Follow-up | 5 | 2 | 1 | 2 | 2
Not completed — Withdrawal by Subject | 3 | 0 | 4 | 5 | 0
Not completed — Vaccine Not Administered | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on enrolled set which includes all participants who have a signed ICF and were assigned to a group, vaccinated, or had an immunogenicity blood draw.
Groups:
- Total: Total of all reporting groups
Arm/Group | CV2CoV Dose Cohort 1 (Group 1a 2µg) | CV2CoV Dose Cohort 1 (Group 1b 4µg) | CV2CoV Dose Cohort 2 (8 µg) | CV2CoV Dose Cohort 3 (12 µg) | CV2CoV Dose Cohort 4 (16 µg) | Total
Number analyzed (Participants) | 24 | 23 | 20 | 21 | 11 | 99
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.5 (15.46) | 44.8 (14.87) | 43.9 (15.77) | 39.7 (12.37) | 37.6 (10.69) | 42.2 (14.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 10 | 8 | 10 | 3 | 48
  Male | 7 | 13 | 12 | 11 | 8 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 11 | 15 | 5 | 47
  Not Hispanic or Latino | 16 | 15 | 9 | 6 | 5 | 51
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs) From Study Vaccination Through the End of the Study
Description: An AESI (serious or nonserious) is defined as an AE or SAE of scientific and medical concern specific to the sponsor's product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor could be appropriate.
Time Frame: From Day 1 up to Day 180 (including Day 180)
Population: Analysis was performed on the Safety set which excludes the participant who attended the visit on Day 1 but was not dosed.
Measure: Count of Participants; unit: Participants
Arm/Group | CV2CoV Dose Cohort 1 (Group 1a 2µg) | CV2CoV Dose Cohort 1 (Group 1b 4µg) | CV2CoV Dose Cohort 2 (8 µg) | CV2CoV Dose Cohort 3 (12 µg) | CV2CoV Dose Cohort 4 (16 µg)
Number analyzed (Participants) | 24 | 22 | 20 | 21 | 11
Participants | 1 | 3 | 2 | 0 | 0

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) From Study Vaccination Through the End of the Study
Description: An SAE is defined as any event that: • Results in death • Is immediately life-threatening • Requires inpatient hospitalization or prolongation of existing hospitalization • Results in persistent or significant disability/incapacity • Is a congenital anomaly/birth defect • Is a spontaneous miscarriage Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered SAEs when, based upon appropriate medical judgment, they may jeopardize the participant or may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.
Time Frame: From Day 1 up to Day 180 (including Day 180)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CV2CoV Dose Cohort 1 (Group 1a 2µg) | CV2CoV Dose Cohort 1 (Group 1b 4µg) | CV2CoV Dose Cohort 2 (8 µg) | CV2CoV Dose Cohort 3 (12 µg) | CV2CoV Dose Cohort 4 (16 µg)
Number analyzed (Participants) | 24 | 22 | 20 | 21 | 11
Participants | 0 | 2 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Medically Attended Adverse Events (MAAEs) From Study Vaccination Through the End of the Study
Description: An MAAE is defined as an AE that results in a visit to a medical professional. Medically attended visits are defined as a telemedicine visit, physician's office visit, urgent care visit, emergency room visit, hospitalization, or death.
Time Frame: From Day 1 up to Day 180 (including Day 180)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CV2CoV Dose Cohort 1 (Group 1a 2µg) | CV2CoV Dose Cohort 1 (Group 1b 4µg) | CV2CoV Dose Cohort 2 (8 µg) | CV2CoV Dose Cohort 3 (12 µg) | CV2CoV Dose Cohort 4 (16 µg)
Number analyzed (Participants) | 24 | 22 | 20 | 21 | 11
Participants | 3 | 4 | 0 | 1 | 1

4. Primary Outcome: Number of Participants With Solicited Local Adverse Events (AEs) up to 7 Days After Study Vaccination
Description: Assessed solicited local reactions were injection site pain, redness, swelling, and lymphadenopathy.
Time Frame: From Day 1 to Day 7 (including Day 7)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CV2CoV Dose Cohort 1 (Group 1a 2µg) | CV2CoV Dose Cohort 1 (Group 1b 4µg) | CV2CoV Dose Cohort 2 (8 µg) | CV2CoV Dose Cohort 3 (12 µg) | CV2CoV Dose Cohort 4 (16 µg)
Number analyzed (Participants) | 24 | 22 | 20 | 21 | 11
Participants
  Injection Site Pain | 7 | 11 | 10 | 13 | 7
  Swelling | 0 | 0 | 1 | 1 | 1
  Redness | 0 | 2 | 0 | 0 | 0
  Lymphadenopathy | 1 | 3 | 2 | 2 | 1

5. Primary Outcome: Number of Participants With Each Solicited Systemic AEs up to 7 Days After Study Vaccination
Description: Assessed solicited systemic reactions were fever, headache, fatigue, myalgia, arthralgia, and chills.
Time Frame: From Day 1 to Day 7 (including Day 7)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CV2CoV Dose Cohort 1 (Group 1a 2µg) | CV2CoV Dose Cohort 1 (Group 1b 4µg) | CV2CoV Dose Cohort 2 (8 µg) | CV2CoV Dose Cohort 3 (12 µg) | CV2CoV Dose Cohort 4 (16 µg)
Number analyzed (Participants) | 24 | 22 | 20 | 21 | 11
Participants
  Fever | 0 | 0 | 1 | 3 | 3
  Myalgia | 6 | 12 | 10 | 12 | 7
  Chills | 3 | 4 | 7 | 10 | 8
  Fatigue | 11 | 9 | 7 | 10 | 5
  Headache | 12 | 7 | 10 | 14 | 7
  Arthralgia | 2 | 5 | 4 | 7 | 2

6. Primary Outcome: Number of Participants With Unsolicited AEs up to 28 Days After Study Vaccination, Including Clinically Relevant Abnormal Clinical Safety Laboratory Findings
Description: An unsolicited AE is defined as any AE that is volunteered from the participant and occurs within 28 days after vaccination.
Time Frame: From Day 1 to Day 28 (including Day 28)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CV2CoV Dose Cohort 1 (Group 1a 2µg) | CV2CoV Dose Cohort 1 (Group 1b 4µg) | CV2CoV Dose Cohort 2 (8 µg) | CV2CoV Dose Cohort 3 (12 µg) | CV2CoV Dose Cohort 4 (16 µg)
Number analyzed (Participants) | 24 | 22 | 20 | 21 | 11
Participants | 4 | 4 | 5 | 5 | 0

7. Secondary Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibody Titers Against Pseudovirus Bearing Spike Protein From SARS CoV 2 Wild Type (WT)
Time Frame: At Day 1, Day 8, Day 15, Day 29, Day 85, and Day 180
Population: The Per Protocol set included all eligible participants who received a dose of study intervention per protocol and who have values at specific timepoint for neutralizing Ab titers against pseudovirus bearing S protein from WT SARS-CoV-2.
Measure: Geometric Mean (Standard Deviation); unit: Titers
Arm/Group | CV2CoV Dose Cohort 1 (Group 1a 2µg) | CV2CoV Dose Cohort 1 (Group 1b 4µg) | CV2CoV Dose Cohort 2 (8 µg) | CV2CoV Dose Cohort 3 (12 µg) | CV2CoV Dose Cohort 4 (16 µg)
Number analyzed (Participants) | 19 | 19 | 13 | 15 | 7
Titers
  Day 1 | 1254.1 (5.54) | 757.7 (8.22) | 1889.5 (3.79) | 1696.6 (2.99) | 1534.3 (2.04)
  Day 8: number analyzed (Participants) | 19 | 16 | 10 | 15 | 6
  Day 8 | 1639.9 (3.72) | 1342.1 (5.49) | 2378.5 (3.15) | 2865.5 (2.43) | 3242.6 (2.22)
  Day 15: number analyzed (Participants) | 19 | 17 | 7 | 14 | 7
  Day 15 | 1801.1 (3.14) | 1651.9 (3.58) | 3316.1 (1.86) | 3372.1 (2.15) | 2395.3 (2.08)
  Day 29: number analyzed (Participants) | 19 | 19 | 11 | 15 | 7
  Day 29 | 2029.9 (3.03) | 1784.3 (3.40) | 3614.7 (2.29) | 3330.6 (2.21) | 2748.7 (1.89)
  Day 85: number analyzed (Participants) | 10 | 14 | 9 | 9 | 5
  Day 85 | 2474.1 (3.24) | 3152.2 (2.73) | 3496.0 (2.16) | 2564.0 (2.26) | 2255.2 (1.84)
  Day 180: number analyzed (Participants) | 10 | 11 | 9 | 10 | 5
  Day 180 | 2231.3 (2.59) | 2206.0 (3.88) | 4025.5 (1.99) | 3045.5 (2.82) | 2356.5 (1.81)

8. Secondary Outcome: Percentage of Participants With Seroresponse (>= 4 Fold Rise From Baseline) at Day 29 After the Booster Dose
Description: Percentage of participants with seroresponse against antigen SARS-CoV-2 WT, Beta, Omicron BA.1, Omicron BA.2, Delta assessed were reported. Seroresponse was defined as greater than equal to (>=) 4-fold increase from Day 1 (Baseline) to the Day 29. The fold rise was calculated as the ratio of the post-vaccination Neutralizing Antibody Titers to the pre-vaccination Neutralizing Antibody Titers.
Time Frame: At Day 29 (29 days post booster dose)
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | CV2CoV Dose Cohort 1 (Group 1a 2µg) | CV2CoV Dose Cohort 1 (Group 1b 4µg) | CV2CoV Dose Cohort 2 (8 µg) | CV2CoV Dose Cohort 3 (12 µg) | CV2CoV Dose Cohort 4 (16 µg)
Number analyzed (Participants) | 19 | 19 | 11 | 15 | 7
Percentage of participants
  WT | 15.8 | 31.6 | 9.1 | 13.3 | 14.3
  Beta | 10.5 | 31.6 | 9.1 | 20.0 | 0.0
  Omicron BA.1 | 15.8 | 21.1 | 9.1 | 20.0 | 0.0
  Omicron BA.2 | 21.1 | 26.3 | 9.1 | 26.7 | 0.0
  Delta | 21.1 | 31.6 | 9.1 | 20.0 | 0.0

9. Secondary Outcome: Geometric Mean Increase (GMI) From Baseline of Neutralizing Antibody Titers Against Pseudovirus Bearing Spike Protein From SARS CoV 2 WT at Each Collection Time Point
Time Frame: At Day 8, Day 15, Day 29, Day 85, and Day 180
Population: as for outcome 7
Measure: Geometric Mean (Standard Deviation); unit: Titers
Arm/Group | CV2CoV Dose Cohort 1 (Group 1a 2µg) | CV2CoV Dose Cohort 1 (Group 1b 4µg) | CV2CoV Dose Cohort 2 (8 µg) | CV2CoV Dose Cohort 3 (12 µg) | CV2CoV Dose Cohort 4 (16 µg)
Number analyzed (Participants) | 19 | 19 | 13 | 15 | 7
Titers
  Day 8: number analyzed (Participants) | 19 | 16 | 10 | 15 | 6
  Day 8 | 1.31 (1.960) | 1.52 (2.068) | 1.30 (1.631) | 1.69 (2.003) | 1.83 (1.725)
  Day 15: number analyzed (Participants) | 19 | 17 | 7 | 14 | 7
  Day 15 | 1.44 (2.048) | 2.35 (3.197) | 1.68 (2.380) | 1.95 (2.300) | 1.56 (1.569)
  Day 29: number analyzed (Participants) | 19 | 19 | 11 | 15 | 7
  Day 29 | 1.62 (2.541) | 2.35 (3.410) | 1.31 (1.872) | 1.96 (2.183) | 1.79 (1.969)
  Day 85: number analyzed (Participants) | 10 | 14 | 9 | 9 | 5
  Day 85 | 1.46 (2.318) | 2.07 (3.429) | 1.15 (2.086) | 1.33 (1.976) | 1.08 (1.429)
  Day 180: number analyzed (Participants) | 10 | 11 | 9 | 10 | 5
  Day 180 | 0.85 (2.128) | 1.67 (2.903) | 1.48 (1.955) | 1.44 (1.765) | 1.13 (1.893)

10. Secondary Outcome: GMTs of Binding Immunoglobulin G (IgG) Against SARS CoV-2 S Protein and Receptor-Binding Domain (RBD)
Time Frame: At Day 8, Day 15, Day 29, Day 85 and Day 180
Population: as for outcome 7
Measure: Geometric Mean (Standard Deviation); unit: Titers
Groups:
- CV2CoV Dose Cohort 4 (16 µg): 8Participants received 16 µg CV2CoV intramuscularly.
Arm/Group | CV2CoV Dose Cohort 1 (Group 1a 2µg) | CV2CoV Dose Cohort 1 (Group 1b 4µg) | CV2CoV Dose Cohort 2 (8 µg) | CV2CoV Dose Cohort 3 (12 µg) | CV2CoV Dose Cohort 4 (16 µg)
Number analyzed (Participants) | 19 | 19 | 13 | 15 | 7
Titers
  Day 8: number analyzed (Participants) | 19 | 16 | 10 | 15 | 6
  Day 8 | 85721.0 (4.00) | 63602.3 (3.55) | 100471.0 (2.66) | 139859.4 (1.88) | 163686.8 (2.14)
  Day 15: number analyzed (Participants) | 19 | 16 | 7 | 14 | 7
  Day 15 | 103076.4 (3.36) | 80210.9 (2.24) | 132016.5 (2.80) | 172621.3 (1.65) | 167769.4 (1.99)
  Day 29: number analyzed (Participants) | 19 | 19 | 11 | 15 | 7
  Day 29 | 103702.2 (3.23) | 101635.2 (2.34) | 137232.9 (2.49) | 136088.9 (1.86) | 112702.8 (2.12)
  Day 85: number analyzed (Participants) | 8 | 14 | 8 | 9 | 4
  Day 85 | 171980.7 (2.57) | 120609.1 (2.73) | 121543.7 (2.92) | 63229.7 (2.15) | 110797.5 (1.51)
  Day 180: number analyzed (Participants) | 8 | 9 | 8 | 10 | 4
  Day 180 | 76009.5 (2.58) | 70208.3 (3.58) | 140651.1 (2.42) | 101287.9 (2.02) | 96157.6 (1.78)

11. Secondary Outcome: GMI From Baseline of Binding IgG Against SARS CoV-2 S Protein and RBD
Time Frame: At Day 8, Day 15, Day 29, Day 85, and Day 180
Population: as for outcome 7
Measure: Geometric Mean (Standard Deviation); unit: Titers
Arm/Group | CV2CoV Dose Cohort 1 (Group 1a 2µg) | CV2CoV Dose Cohort 1 (Group 1b 4µg) | CV2CoV Dose Cohort 2 (8 µg) | CV2CoV Dose Cohort 3 (12 µg) | CV2CoV Dose Cohort 4 (16 µg)
Number analyzed (Participants) | 19 | 19 | 13 | 15 | 7
Titers
  Day 8: number analyzed (Participants) | 19 | 16 | 10 | 15 | 6
  Day 8 | 1.32 (1.671) | 1.44 (1.575) | 1.48 (1.859) | 1.57 (1.623) | 1.28 (1.421)
  Day 15: number analyzed (Participants) | 19 | 16 | 7 | 14 | 7
  Day 15 | 1.58 (2.181) | 2.51 (2.936) | 1.62 (2.107) | 1.88 (1.856) | 1.44 (1.435)
  Day 29: number analyzed (Participants) | 19 | 19 | 11 | 15 | 7
  Day 29 | 1.59 (2.711) | 2.48 (2.990) | 1.29 (1.530) | 1.53 (1.741) | 0.96 (1.345)
  Day 85: number analyzed (Participants) | 8 | 14 | 8 | 9 | 4
  Day 85 | 0.95 (1.317) | 1.88 (3.111) | 1.34 (2.730) | 0.71 (1.732) | 0.71 (1.417)
  Day 180: number analyzed (Participants) | 8 | 9 | 8 | 10 | 4
  Day 180 | 0.78 (1.801) | 1.52 (3.789) | 1.38 (1.938) | 1.18 (1.711) | 0.62 (2.535)

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs) were collected through the entire period of the study (from Day 1 up to study end [Day 180]). Solicited adverse events were collected from Day 1-7, unsolicited adverse events from Day 1-30, Abnormal Clinical Safety Laboratory Findings from Day 1-28, Non-Serious Covid-19 Adverse Events from Day 1 up to Study End [Day 180] after Study Vaccination
Description: Adverse events were assessed in safety set which exclude participant who attended the visit on Day 1 but was not dosed.
Arm/Group | CV2CoV Dose Cohort 1 (Group 1a 2µg) | CV2CoV Dose Cohort 1 (Group 1b 4µg) | CV2CoV Dose Cohort 2 (8 µg) | CV2CoV Dose Cohort 3 (12 µg) | CV2CoV Dose Cohort 4 (16 µg)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/22 | 0/20 | 0/21 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/24 | 2/22 | 0/20 | 0/21 | 0/11
Other Adverse Events (participants affected / at risk) | 18/24 | 17/22 | 16/20 | 18/21 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CV2CoV Dose Cohort 1 (Group 1a 2µg) (N=24) | CV2CoV Dose Cohort 1 (Group 1b 4µg) (N=22) | CV2CoV Dose Cohort 2 (8 µg) (N=20) | CV2CoV Dose Cohort 3 (12 µg) (N=21) | CV2CoV Dose Cohort 4 (16 µg) (N=11)
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CV2CoV Dose Cohort 1 (Group 1a 2µg) (N=24) | CV2CoV Dose Cohort 1 (Group 1b 4µg) (N=22) | CV2CoV Dose Cohort 2 (8 µg) (N=20) | CV2CoV Dose Cohort 3 (12 µg) (N=21) | CV2CoV Dose Cohort 4 (16 µg) (N=11)
Injection site pain (General disorders) | 7 | 11 | 10 | 13 | 7
Fatigue (General disorders) | 11 | 9 | 7 | 10 | 5
Chills (General disorders) | 3 | 4 | 7 | 10 | 8
Fever (General disorders) | 0 | 0 | 1 | 3 | 3
Injection site swelling (General disorders) | 0 | 0 | 1 | 1 | 1
Injection site erythema (General disorders) | 0 | 2 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0
Injection site bruising (General disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 12 | 7 | 10 | 14 | 7
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 12 | 10 | 12 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 5 | 4 | 8 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 3 | 2 | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 1 | 3 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/37/NCT05260437/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT05260437/SAP_001.pdf